CLINICAL TRIAL: NCT00781833
Title: Case Study Testing the Use of Implanted Microstimulators for Decreasing Spasticity and Improving Motion Following Spinal Cord Injury
Brief Title: Use of Implanted Microstimulators for Decreasing Spasticity and Improving Motion Following Spinal Cord Injury
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Participation of single subject enrolled was terminated.
Sponsor: The Alfred E. Mann Foundation for Scientific Research (Other)
Collaborators: Walter Reed Army Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMF CP-005
Record Dates: First submitted 2008-10-27; First posted 2008-10-29 (Estimated); Last update posted 2012-01-23 (Estimated); Status verified 2012-01

CONDITIONS: Spinal Cord Injury at C5-C7 Level With Incomplete Lesion
Keywords: Therapeutic Electric Stimulation; Functional Electric Stimulation; Implantable Stimulator; Muscle Strength; Muscle Spasticity
MeSH Terms: conditions — Muscle Spasticity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Intramuscular Electrical Stimulation
  Interventions: Device: Radio Frequency Microstimulator

INTERVENTIONS:
Device: Radio Frequency Microstimulator — Implantable peripheral muscle microstimulator, delivering controlled pulsatile stimulation to femoral nerves for knee extension and peroneal nerves for dorsiflexion.

SUMMARY:
The primary aims of this study are to determine the safety of the RFM System (Alfred Mann Foundation, Santa Clarita, CA) in a patient with incomplete SCI and the effect of the RFM system on lower limb strength and spasticity. The secondary aim is to analyze any improvement in the participant's mobility.

DETAILED DESCRIPTION:
Restoring mobility after spinal cord injury (SCI) is one of the most important goals of rehabilitation. Even for patients with partial lower limb motor function after SCI, many have limited mobility because of significant spasticity. Therapeutic electrical neuromuscular stimulation (TNS) has been used to improve muscle tone and strength and to enable walking and standing in patients with SCI. We propose to use the Radio Frequency Microstimulator (RFM) System, a new and novel implantable TNS system developed by the Alfred E. Mann Foundation, to improve muscle strength and reduce spasticity in a patient with incomplete SCI. The RFM System has several advantages over current TNS systems. The RFM implant devices are small enough (diameter 2.4 mm, length 16.7 mm) to be inserted using an incision approximately 5 mm long and have no lead wires passing through the skin since the microstimulator contains both the anode and cathode. Implanted RFM devices can be placed near multiple motor points and/or nerves and are controlled individually using radio frequency technology. Up to six (6) RFM devices will be inserted, two to three in each lower limb to provide stimulation to a patient's bilateral knee extensors (femoral nerve stimulation) and ankle dorsiflexors (peroneal nerve stimulation) to assess the effects on muscle strength, limb spasticity and patient mobility.

ELIGIBILITY:
Inclusion Criteria:

* an incomplete C6 ASIA C (Central Cord) spinal cord injury
* lower motor function impaired and suffers from significant spasticity (Ashworth scale 4)
* able to ambulate approximately 10-20 feet with a rolling walker and minimal assistance
* has sufficient endurance to complete at least two 20-minute therapy sessions per day
* cognitive abilities are intact

Exclusion Criteria:

* psychiatric diagnosis
* medical contraindications
* history of bleeding disorders
* allergy to anesthesia
* acute or progressive disease
* active implantable device

Ages: 55 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2008-10; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Throughout
Lower Limb Strength | 6, 12, 24 weeks, 12, 24 months
Lower Limb Spasticity | 6, 12, 24 weeks, 12, 24 months

SECONDARY OUTCOMES:
Mobility | 6, 12, 24 weeks, 12, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: KEVIN F FITZPATRICK, M.D., Principal Investigator — Walter Reed Army Medical Center
Locations (1):
- Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States